CLINICAL TRIAL: NCT01684254
Title: An In-Shoe Device to Monitor Toe-Walking in Children With Cerebral Palsy
Status: Terminated | Type: Observational
Why Stopped: Lack of funding
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: Peabody Foundation, Inc. (Other)
Responsible Party: Principal Investigator, Paolo Bonato, Director, Motion Analysis Laboratory, Spaulding Rehabilitation Hospital
Other Study IDs: 2007-P-000837
Record Dates: First submitted 2012-09-10; First posted 2012-09-12 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Children With Cerebral Palsy
Keywords: Cerebral Palsy; Home monitoring; Gait; Sensorized Shoe
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Children with Cerebral Palsy (CP)

SUMMARY:
The present project will focus on evaluating the technical efficacy of the in-shoe gait monitoring device (ActiveGait) through laboratory based biomechanical gait assessments of children who exhibit gait deviations due to CP or idiopathic toe walking wearing the device.

DETAILED DESCRIPTION:
The investigators on this protocol intend to develop the device and rely on it to propose a Toe Walk Severity (TWS) index, a novel outcome measure for quantifying changes in severity of toe walking over time and for assessing the outcome of surgical and non-surgical interventions.

Tasks include:

A.Validate data acquisition measurements in laboratory setting compared to gold-standard video analysis and field (outside of laboratory).

B.Develop multi-stage classification algorithm from subset of laboratory and field data.

C.Validate classification algorithm against random subsets of laboratory and field data.

D.Explore the development of a Toe Walking Severity (TWS) index from available biomechanical and ActiveGait data for different ambulatory conditions.

E.Perform longitudinal study of the childhood toe walking population including both laboratory analysis and at-home monitoring using ActiveGait technology.

F.Analyze statistically the sensitivity and specificity of the TWS index compared to clinical observations. Gather evidence that the TWS index provides a means to track changes in severity of toe walking over time.

ELIGIBILITY:
Inclusion Criteria:

* able to ambulate 50 feet on level ground without the assistance of a person
* able to ambulate on ramps and stairs without the assistance of a person
* demonstrate a toe-walking pattern at the time of enrollment
* medically stable
* able to understand directions and follow simple instructions

Exclusion Criteria:

* any cardiopulmonary, orthopedic, and neurological conditions other than CP that would prevent them from performing the motor tasks of interest

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children diagnosed with CP
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2010-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Toe Walking Severity (TWS) index | 1 day
  Measure for quantifying changes in severity of toe walking over time based on Center of Pressure trajectories computed by the sensorized insole

SECONDARY OUTCOMES:
Edinburgh Visual Scale (EVS) score | 1 day
  Clinical measure of severity of gait deviation

CONTACTS AND LOCATIONS:
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States